CLINICAL TRIAL: NCT05965960
Title: Investigating Local Field Potential Correlates of Transcranial Ultrasound Stimulation in Patients With Movement Disorders
Brief Title: Investigating LFP Correlates of TUS in Patients With Movement Disorders
Acronym: TUS-LFP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 20-5740#2
Record Dates: First submitted 2023-06-07; First posted 2023-07-28 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease; Essential Tremor; Dystonia
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Dystonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The subject will be blind to stimulation condition (sham/active TUS). The assessor will be blind to stimulation condition (sham/active TUS) while analyzing LFPs. The UPDRS examination will be video-recorded and blindly assessed by a research team member.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Low Intensity Transcranial Focused Ultrasound (Active Comparator): NeuroFUS device stimulation with 4 channel transducer Stimulation target = M1/GPi Stimulation parameters = Theta burst protocol and 30 Watts
  Interventions: Device: TUS Active
- Sham Low Intensity Transcranial Focused Ultrasound (Sham Comparator): NeuroFUS device stimulation with 4 channel transducer Stimulation target = M1/GPi Stimulation parameters = Theta burst protocol and 0 Watts
  Interventions: Device: TUS Sham

INTERVENTIONS:
Device: TUS Active — Bilateral M1s/GPis will be sonicated using NeuroFUS device for two minutes per hemisphere with theta burst protocol and 30 W/cm2 Isppa
  Arms: Active Low Intensity Transcranial Focused Ultrasound
Device: TUS Sham — Bilateral M1s/GPis will be sonicated using NeuroFUS device for two minutes per hemisphere with theta burst protocol and 0 W/cm2 Isppa
  Arms: Sham Low Intensity Transcranial Focused Ultrasound

SUMMARY:
Transcranial Ultrasound Stimulation (TUS) is an emerging non-invasive brain stimulation(NIBS) technique that can be used on both superficial and deep brain targets with a high spatial resolution as small as a few cubic millimeters. Neural correlates of TUS have yet been elucidated. To date, no intracranial recordings (i.e., local field potential [LFP]) have been captured during or after TUS in patients with movement disorders. In this study, we are aiming to profile basal ganglia LFP activity during and after TUS by using a DBS system that is capable of recording LFP. This can shed light on mechanisms of TUS, as well as allow identification of a neurophysiological biomarker that can be used to tune the TUS sonication parameters for future clinical trials.

DETAILED DESCRIPTION:
Experiment 1: Subjects will be randomly assigned to either the sham or active stimulation group during the first study visit. In the second study visit, there will be a crossover between the groups, with all subjects undergoing one sham and one active stimulation visit before the study is completed. During the active stimulation visit, a theta burst protocol (Isppa: 30 W/cm2, burst length: 20 ms, period: 200 ms, frequency 500 kHz) will be used to sonicate the bilateral primary motor cortices (M1) or globus pallidus interna (GPi) for 2 minutes. The sham group involves sonications performed with the power set to 0 watts over bilateral M1s/GPis. In both groups, the subjects will be masked using white noise transmitted through earbuds. The targets will be identified anatomically using structural MRIs and a neuronavigation system.

The Percept PC DBS system will be used to record local field potentials (LFPs) from the subthalamic nucleus (STN) or globus pallidus internus (GPI) at various time points: before (baseline) and during the sonications, as well as at 10-, 30-, and 45-minute intervals after the sonications. These recordings will be obtained while the subjects engage in a finger tapping task monitored by an accelerometer, as well as during resting periods. The power of LFPs across different frequencies will be compared and correlated with the velocity observed during the finger tapping task.

Following the completion of sham and active stimulation visits, the subjects will have the opportunity to participate in an optional control group visit, which entails sonication of the occipital cortex utilizing the theta burst protocol.

Experiment 2: TUS will be utilized to target the area directly over the DBS lead, while concurrently recording LFPs to identify any stimulation artifact indicative of target area-sonication engagement.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with movement disorders (diagnosed by a movement disorder specialist)
2. Implantation of a Percept PC DBS system at least one month before the sonications
3. Stable dopaminergic medication dose for a minimum of 4 weeks

Exclusion Criteria:

1. Concomitant neurological conditions (stroke, seizure, dementia, major depression / psychiatric disorders, active drug abuse/addiction and major neuromuscular/musculoskeletal diseases)
2. Declined cognitive scores (MoCA score < 22)
3. Implants (cardiac pacemaker, implantable cardioverter-defibrillator, intracranial devices other than DBS system such as shunts and MR-unsafe devices)
4. History of intracranial lesioning procedures
5. Major systemic illness, infection or pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
LFP power (Experiment 1) | 5 minutes long recordings during both study visits at 1) Baseline (20-30 minutes before sonication), 2) during sonication, 3) 10 minutes after sonication, 4) 30 minutes after sonication, and 5) 45 minutes after sonication
  The change of power of LFPs across different frequencies
Stimulation artifact (Experiment 2) | Online during sonications
  Presence of a stimulation artifact during LFP recordings

SECONDARY OUTCOMES:
UPDRS (Experiment 1) | Two assessments will be conducted during each study visit: one at baseline (within the first minute of the study) and the other upon completion of the study visit (between 120 and 130 minutes after the study visit initiation).
  Change of UPDRS score
Finger tapping task (Experiment 1) | LFPs during finger tapping will be recorded at each visit for half minute at 1) Baseline (20-30 minutes before sonication), 2) 10 minutes after sonication, 3) 30 minutes after sonication, and 4) 45 minutes after sonication
  Correlation of LFP power change with the velocity change during finger tapping task as recorded by an accelerometer
Adverse effect profile (Experiment 1 and 2) | From the initiation of the study up to 1 day after its completion.
  Presence of adverse effects as reported subjectively by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Robert Chen, MBBS, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No